CLINICAL TRIAL: NCT05764265
Title: An Open-label Extension Study to Investigate Efficacy, Safety and Tolerability of LTP001 in Participants With Pulmonary Arterial Hypertension
Brief Title: Extension Study of Efficacy and Safety of LTP001 in Pulmonary Arterial Hypertension Participants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTP001A12201E1; 2022-002007-38 (EudraCT Number)
Record Dates: First submitted 2023-01-10; First posted 2023-03-10 (Actual); Results first posted 2025-12-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LTP001 (Experimental): Participants received LTP001, 6 mg, orally once daily in the morning for approximately 39 weeks
  Interventions: Drug: LTP001

INTERVENTIONS:
Drug: LTP001 — LTP001, 6 mg, was administered orally once daily in the morning

SUMMARY:
The purpose of this study was to measure the long-term safety and efficacy profile of LTP001 in participants with pulmonary arterial hypertension (PAH). The study offered participants who had completed the CLTP001A12201 double-blind parent study in PAH an opportunity to receive LTP001 (whether they were on LTP001 or not). Unblinding of the treatment received in CLTP001A12201 was generally not needed but could occur on request by the investigator.

DETAILED DESCRIPTION:
This was a non-randomized, open-label extension study of LTP001 for participants with PAH who completed the parent Study CLTP001A12201. Eligible participants were presented with the opportunity to enroll in the extension study at the end of treatment visit of the parent study. Participants in the extension study were planned to receive a once-daily dose of LTP001 for 52 weeks regardless of their parent study treatment (i.e. LTP001 or placebo). The study duration was planned up to 54 weeks with a treatment duration up to 52 weeks and maximum 2-week transition period from the CLTP001A12201 study. The visit frequency was planned to include visits at Weeks 1, 5, 13, 26, 39, 52, and 54 along with optional visits at the discretion of the Investigators at Weeks 9 and 17.

Due to the study termination, no patient reached Week 52. After the termination announcement, following the instruction to immediately stop treatment for all participants, an end-of-treatment (EOT) visit was conducted. Sites were advised to complete protocol-required assessments based on investigator judgement and patient willingness to undergo procedures, with a primary focus on ensuring a safe exit from the study. Most sites performed only a few safety assessments, and only a minimal number of patients completed an echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must have been obtained before any assessment was performed.
* Participant was currently completing the Novartis-sponsored study CLTP001A12201 in PAH and completed key efficacy and safety procedures up to the end of treatment of the core study, without meeting discontinuation criteria in the core study.
* Willingness and ability to comply with scheduled visits, treatment plans and any other study procedures.
* In the opinion of the Investigator would benefit from LTP001 treatment.

Exclusion Criteria:

* History of hypersensitivity to the study treatment.
* Sexually active males not committing to condom use precautions: sexually active males must have used a condom during intercourse while taking drug and for 24 hours after stopping study medication and should not father a child in this period nor donate sperm. A condom was required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
* Required or planned transplant or heart/lung surgery.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they were using highly effective methods of contraception while taking study treatment and until EOT visit (2 weeks post-last treatment). Highly effective contraception methods included:
* Total abstinence (when this was in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal were not acceptable methods of contraception.
* Female sterilization (had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman had been confirmed by follow up hormone level assessment.
* Male sterilization (at least 6 months prior to screening). For female participants on the study, the vasectomized male partner should have been the sole partner for that participant
* Use of oral, estrogen and progesterone, injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.

In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

Women were considered post-menopausal if they had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate history of vasomotor symptoms). Women were considered not of child-bearing potential if they were post-menopausal or had surgical bilateral oophorectomy (with or without hysterectomy) or total hysterectomy at least six weeks prior. In the case of oophorectomy alone, only when the reproductive status of the woman had been confirmed by follow up hormone level assessment was she considered not of child bearing potential.

* Pregnant or nursing (lactating) women, where pregnancy was defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Acute or chronic impairment (other than dyspnea), which would limit the ability to comply with study requirements, including interference with physical activity or execution of study procedures such as 6MWT (e.g., angina pectoris, claudication, musculoskeletal disorder, need for walking aids).
* Permanent discontinuation of Novartis drug in the core efficacy study due to toxicity or disease progression despite active treatment, non-compliance to study procedures, withdrawal of consent or any other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Pulmonary Associates PA, Mesa, Arizona, United States
- Novartis Investigative Site, Caba, Buenos Aires, Argentina
- Germany (2):
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Heidelberg
- Novartis Investigative Site, Amsterdam, North Holland, Netherlands
- Poland (3):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Wroclaw
- Spain (3):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
- Novartis Investigative Site, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2605

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 31 participants who completed the parent study up to the end of treatment were screened for the extension study.
Groups:
- LTP001 6 mg (Actual Treatment in CLTP001A12201): Participants had received LTP001, 6 mg, in Study CLTP001A12201, and continued to receive LTP001, 6 mg, orally once daily in the morning for approximately 39 weeks in this extension study
- LTP001 6 mg (Placebo in CLTP001A12201): Participants had received placebo in Study CLTP001A12201, followed by LTP001, 6 mg, orally once daily in the morning for approximately 39 weeks in this extension study
Period: Overall Study
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Started | 23 | 8
Completed | 0 | 0
Not Completed | 23 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 8
Not completed — Study Terminated By Sponsor | 20 | 0
Not completed — Participant Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201) | Total
Number analyzed (Participants) | 23 | 8 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.0 (11.76) | 48.4 (13.35) | 47.4 (11.97)
Age, Customized [Number; unit: Participants]
  18 - <65 | 20 | 7 | 27
  65 - <85 | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 6 | 27
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 21 | 7 | 28
  American Indian or Alaskan | 2 | 0 | 2
  Asian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Incidence and severity of adverse events (AEs) by treatment group, including changes in the vital signs, electrocardiogram and laboratory results qualifying and reported as AEs. Due to the study termination, no patient reached Week 52. At the end of treatment visit, final safety assessments were performed.
Time Frame: Up to approximately 45 weeks
Population: The safety analysis set included all participants who received any study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 23 | 8
Percentage of participants
  AEs | 52.2 | 62.5
  Serious AEs | 17.4 | 0

2. Secondary Outcome: Change From Baseline in Average Cardiac Output (CO) at Week 26
Description: Right heart catheterization (RHC) assessment was performed to assess several hemodynamic variables in pulmonary hypertension, including CO.
Time Frame: Baseline, Week 26
Population: The pharmacodynamic (PD) analysis set included all participants who received study treatment and had no protocol deviations with a relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 6 | 2
liters per minute | -0.111 (0.2153) | -0.065 (0.5916)

3. Secondary Outcome: Change From Baseline in Mean Pulmonary Artery (PA) Pressure at Week 26
Description: Right heart catheterization (RHC) assessment was performed to assess several hemodynamic variables in pulmonary hypertension, including PA pressure.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 6 | 2
mmHg | 3.8 (8.18) | -1.5 (7.78)

4. Secondary Outcome: Change From Baseline in Pulmonary Capillary Wedge Pressure (PCWP) at Week 26
Description: Right heart catheterization (RHC) assessment was performed to assess several hemodynamic variables in pulmonary hypertension, including pulmonary capillary wedge pressure (PCWP).
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 6 | 2
mmHg | -1.0 (1.79) | -0.5 (0.71)

5. Secondary Outcome: Change From Baseline in Right Heart Catheterization Pulmonary Vascular Resistance (PVR) at Week 26
Description: PVR was defined as the resistance against blood flow from the pulmonary artery to the left atrium measured in dynes.sec.cm-5.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dynes.sec.cm-5
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 6 | 2
dynes.sec.cm-5 | 100.058 (95.5879) | -7.445 (34.8250)

6. Secondary Outcome: Change From Baseline in Right Atrium (RA) Pressures at Week 26
Description: The Right Heart Catheterization (RHC) assessment was performed to assess several hemodynamic variables in pulmonary hypertension, including RA pressures.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 6 | 2
mmHg | -1.5 (6.22) | 0.0 (2.83)

7. Secondary Outcome: Change From Baseline in Systemic Vascular Resistance (SVR) at Week 26
Description: The Right Heart Catheterization (RHC) assessment was performed to assess several hemodynamic variables in pulmonary hypertension, including SVR.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dynes.sec.cm-5
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 6 | 2
dynes.sec.cm-5 | 166.748 (128.6202) | -49.710 (28.5388)

8. Secondary Outcome: Change From Baseline in Six Minute Walk Distance (6MWD)
Description: 6MWD test measures the distance that a participant can walk on a flat, hard surface in a period of 6 minutes. Due to the study termination, no patient reached Week 52. At the end of treatment (EOT) visit, final safety assessments were performed based on investigator judgement and patient willingness to undergo procedures.
Time Frame: Baseline, Week 26, up to 39 weeks (EOT)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 16 | 2
meters
  Week 26 n=6,2: number analyzed (Participants) | 6 | 2
  Week 26 n=6,2 | -33.7 (55.60) | -9.0 (25.46)
  EOT n=16,2 | -6.3 (50.21) | -1.0 (1.41)

9. Secondary Outcome: Change From Baseline in Tricuspid Annular Plane Systolic Excursion (TAPSE)
Description: Key right ventricular (RV) function endpoints such as tricuspid annular plane systolic excursion (TAPSE) were assessed with echocardiography. Due to the study termination, no patient reached Week 52. At the end of treatment (EOT) visit, final safety assessments were performed based on investigator judgement and patient willingness to undergo procedures. Only a minimal number of patients completed an echocardiogram (Echo).
Time Frame: Baseline, Week 26, up to 39 weeks (EOT)
Population: The pharmacodynamic (PD) analysis set included all participants who received study treatment and had no protocol deviations with a relevant impact on PD data. Number analyzed is the number of participants with data available at the specified time points.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 7 | 2
centimeters
  Week 26 n=6,2: number analyzed (Participants) | 6 | 2
  Week 26 n=6,2 | 0.03 (0.175) | 0.00 (0.283)
  EOT n=7,0: number analyzed (Participants) | 7 | 0
  EOT n=7,0 | 0.01 (0.682) |

10. Secondary Outcome: Change From Baseline in Tricuspid Annular Plane Systolic Velocity (TASV)
Description: Key right ventricular (RV) function endpoints such as tricuspid annular systolic velocity (TASV) were assessed with echocardiography. Due to the study termination, no patient reached Week 52. At the end of treatment (EOT) visit, final safety assessments were performed based on investigator judgement and patient willingness to undergo procedures. Only a minimal number of patients completed an echocardiogram (Echo).
Time Frame: Baseline, Week 26, up to 39 weeks (EOT)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 7 | 2
centimeters per second
  Week 26 n=6,2: number analyzed (Participants) | 6 | 2
  Week 26 n=6,2 | -2.2 (3.43) | -0.5 (0.71)
  EOT n=7,0: number analyzed (Participants) | 7 | 0
  EOT n=7,0 | -2.6 (1.90) |

11. Secondary Outcome: Change From Baseline in Peak Velocity of Excursion (RV S')
Description: Key right ventricular (RV) function per echocardiography. The terms Tricuspid Annular Systolic Velocity (TASV) and Peak Velocity of Excursion (RV S') are synonymous in echocardiography to describe the peak systolic velocity of the lateral tricuspid annulus. Including both TASV and RV S' as separate secondary endpoints was an oversight in the protocol as the data, calculation, and analyses for both (TASV and RV S') are identical. Therefore, the TASV and RV S' data in this results disclosure are the same. Due to the study termination, no patient reached Week 52. At the end of treatment (EOT) visit, final safety assessments were performed based on investigator judgement and patient willingness to undergo procedures. Only a minimal number of patients completed an echocardiogram (Echo).
Time Frame: Baseline, Week 26, up to 39 weeks (EOT)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 7 | 2
centimeters per second
  Week 26 n=6,2: number analyzed (Participants) | 6 | 2
  Week 26 n=6,2 | -2.2 (3.43) | -0.5 (0.71)
  EOT n=7,0: number analyzed (Participants) | 7 | 0
  EOT n=7,0 | -2.6 (1.90) |

12. Secondary Outcome: Change From Baseline in Fractional Area Change (FAC)
Description: Key right ventricular (RV) function endpoints such as RV fractional area change (RV FAC) were assessed with echocardiography. Due to the study termination, no patient reached Week 52. At the end of treatment (EOT) visit, final safety assessments were performed based on investigator judgement and patient willingness to undergo procedures. Only a minimal number of patients completed an echocardiogram (Echo).
Time Frame: Baseline, Week 26, up to 39 weeks (EOT)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 6 | 1
percent
  Week 26 n=6,1 | -0.87 (6.162) | 7.30 (NA) — Standard deviation was not calculable due to the single data point.
  EOT n=6,0: number analyzed (Participants) | 6 | 0
  EOT n=6,0 | 0.97 (5.290) |

13. Secondary Outcome: Change From Baseline in Quality of Life Measured by the emPHasis-10 Questionnaire
Description: emPHasis-10 is a questionnaire with 10 questions designed to determine how pulmonary hypertension affects a participant's life. Each item is scored on a scale of 0 to 5, with a total score ranging from 0 to 50. A higher score indicates worse quality of life. Due to the study termination, no patient reached Week 52. At the end of treatment (EOT) visit, final safety assessments were performed based on investigator judgement and patient willingness to undergo procedures.
Time Frame: Baseline up to 39 weeks (EOT)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 3 | 1
score | 1.476 (2.3226) | 1.000 (NA) — Standard deviation was not calculable due to the single data point.

14. Secondary Outcome: Change From Baseline in Quality of Life Measured by the PAH-SYMPACT Questionnaire
Description: PAH-SYMPACT is a questionnaire used to assess pulmonary arterial hypertension symptoms and their impact. Individual item scores range from 0 to 4. Total score is calculated as the sum of the scores for the individual items divided by the number of items. A higher score indicates more severe symptoms/impacts. Due to the study termination, no patient reached Week 52. At the end of treatment (EOT) visit, final safety assessments were performed based on investigator judgement and patient willingness to undergo procedures.
Time Frame: Baseline up to 39 weeks (EOT)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 2 | 1
score | 2.929 (2.3234) | -0.833 (NA) — Standard deviation was not calculable due to the single data point.

15. Secondary Outcome: Time to Clinical Worsening
Description: Time to any of the following:
  * Death
  * Hospital stay greater than 24 hours due to worsening of pulmonary arterial hypertension
  * Worsening of PAH resulting in need for lung transplantation or balloon atrial septostomy
  * Initiation of parenteral prostanoid therapy, initiation of oxygen therapy, initiation of any other pulmonary arterial hypertension-specific therapies or need for increase of diuretics for more than 4 weeks due to worsening of pulmonary arterial hypertension
  * Significant drop in six-minute walk distance Due to the study termination, no patient reached Week 52. At the end of treatment (EOT) visit, final safety assessments were performed based on investigator judgement and patient willingness to undergo procedures.
Time Frame: Baseline up to 39 weeks (EOT)
Population: The pharmacodynamic (PD) analysis set included all participants who received study treatment and had no protocol deviations with a relevant impact on PD data. Number analyzed is the number of participants with an event up to and including the end time of the interval.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 6 | 0
days | 346.0 [187.0 to NA] — The upper limit of 95% CI was not calculable due to an insufficient number of participants with events. |

16. Secondary Outcome: Change From Baseline in N-terminal Fragment of the Prohormone B-type Natriuretic Peptide (NT-ProBNP)
Description: NT-proBNP is a blood biomarker to assess right ventricular distress. Due to the study termination, no patient reached Week 52. At the end of treatment (EOT) visit, final safety assessments were performed based on investigator judgement and patient willingness to undergo procedures.
Time Frame: Baseline up to 39 weeks (EOT)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picomoles per liter
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201)
Number analyzed (Participants) | 19 | 6
picomoles per liter | 3.832 (31.2255) | 7.250 (16.6033)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 6 weeks post treatment, up to approximately 45 weeks.
Groups:
- Total: Total
Arm/Group | LTP001 6 mg (Actual Treatment in CLTP001A12201) | LTP001 6 mg (Placebo in CLTP001A12201) | Total
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/8 | 0/31
Serious Adverse Events (participants affected / at risk) | 4/23 | 0/8 | 4/31
Other Adverse Events (participants affected / at risk) | 5/23 | 5/8 | 10/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LTP001 6 mg (Actual Treatment in CLTP001A12201) (N=23) | LTP001 6 mg (Placebo in CLTP001A12201) (N=8) | Total (N=31)
Medical device site haemorrhage (General disorders and administration site conditions) | 1 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 1
Disseminated gonococcal infection (Infections and infestations) | 1 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LTP001 6 mg (Actual Treatment in CLTP001A12201) (N=23) | LTP001 6 mg (Placebo in CLTP001A12201) (N=8) | Total (N=31)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Eczema eyelids (Eye disorders) | 0 | 1 | 1
Fatigue (General disorders and administration site conditions) | 0 | 1 | 1
Bartholinitis (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 3
Tooth abscess (Infections and infestations) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT05764265/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT05764265/SAP_001.pdf